CLINICAL TRIAL: NCT03084848
Title: Cerebral Bases of the Cognitive Learning in the Executive Control In the Adolescence
Brief Title: Executive Training and Brain in Adolescent
Acronym: APEX-ADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D15-P017; 2015-A00811-48 (Other: ANSM)
Record Dates: First submitted 2016-04-06; First posted 2017-03-21 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: brain/cognitive measures; condition; inhibitor control; training at adolescence
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active control (Experimental)
  Interventions: Other: Training
- Inhibitor control (Experimental)
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — 25 training sessions of 15 minutes per day, 5 days a week for a month of crystallised intelligence
  Arms: Active control
Other: Training — 25 training sessions of 15 minutes per day, 5 days a week for a month of inhibitory control
  Arms: Inhibitor control

SUMMARY:
The purpose of this study is to investigate the cognitive and brain effects of inhibitory control (IC) training at adolescence.

DETAILED DESCRIPTION:
Brain imaging now allows to study non-invasively cognitive learning processes. An area of strong scientific interest is the development of executive control, an essential cognitive domain for academic and professional success and for mental and physical health. These functions are essentially located within the prefrontal cortex, characterising by a late maturation until the end of adolescence and, while under genetic control, can likely be improved with targeted interventions. The objective of this project is simple and innovative: testing in adolescents with the most appropriate brain imaging technologies available today (the Magnetic Resonance Imaging, MRI), the effect of an executive training focused on the inhibitory control (IC). This project aims at precisely testing the effect at the cognitive and brain levels of IC training in adolescence. To do this, the investigators will recruit two groups of 30 teenagers aged 16 to 17 years old, each assigned to one of two learning situations: IC vs Active Control (AC). Each participant will participate in 25 training sessions of 15 minutes per day, 5 days a week for a month. Brain structural and functional differences in the brain and between the pre-test and post-test related to intense IC training will be correlated with cognitive progress.

ELIGIBILITY:
Inclusion Criteria:

* 16-17 years old
* girl or boy ;
* French mother tongue;
* Handedness: Right;
* Schooled in a level corresponding to its age (2nd or 1st)
* Informed consent signed by the (s) holder (s) of parental authority, in agreement with the teenager
* Normal medical, neurological, neuroradiological examinations.
* Health insurance

Exclusion Criteria:

* classical exclusion criteria for MRI
* Has chronic use of alcohol or drugs;
* Abuse or substance dependence (excluding nicotine) or a toxic over 5 years or has led to comas (overdoses)
* Cognitive disorders of sudden onset that may reflect a stroke; history of head trauma with loss of consciousness for more than 1 hour, or encephalitis;
* A chronic neurological disorder, psychiatric, endocrine, hepatic and infectious disorder;
* Major disease history (diabetes, chronic lung disease, heart disorder, metabolic, hematologic, endocrine or immunological severe cancer);
* A medication that may interfere with brain imaging measures (psychotropic drugs, hypnotics, anxiolytics, antipsychotics, anti-Parkinson, benzodiazepines, anti-inflammatory drugs, antiepileptics, antihistamines, analgesics and muscle relaxants central);
* dyschromatopsia
* Impossibility to submit itself to the study for geographical or psychiatric reasons;
* Pregnant and lactating women;
* Has pervasive developmental disorders and / or acquisitions identified by parents or legal guardian and (or) the teachers;
* Cerebral palsy;
* Fine motor disorder
* Unaccompanied by parent (s) (s) or at least a person with parental authority during the visit to the research platform;
* Tattoo on the head, neck or shoulders

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Brain plasticity : Longitudinal cortical thickness change | Baseline
Brain plasticity : Longitudinal cortical thickness change | one month IC training

CONTACTS AND LOCATIONS:
Overall Officials: Catherine OPPENHEIM, Principal Investigator — Centre Hospitalier Sainte-Anne; Arnaud Cachia, PhD, Pr, Study Director — University Paris Descartes
Locations (2):
- France (2):
  - Centre de Recherche Clinique (CRC) - CHSA, Paris
  - Centre Hospitalier Sainte-Anne, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahr E, Houde O, Borst G. Inhibition of the mirror generalization process in reading in school-aged children. J Exp Child Psychol. 2016 May;145:157-65. doi: 10.1016/j.jecp.2015.12.009. Epub 2016 Jan 27. PMID 26827098
- [Background] Cachia A, Borst G, Vidal J, Fischer C, Pineau A, Mangin JF, Houde O. The shape of the ACC contributes to cognitive control efficiency in preschoolers. J Cogn Neurosci. 2014 Jan;26(1):96-106. doi: 10.1162/jocn_a_00459. Epub 2013 Aug 5. PMID 23915057
- [Background] Borst G, Cachia A, Vidal J, Simon G, Fischer C, Pineau A, Poirel N, Mangin JF, Houde O. Folding of the anterior cingulate cortex partially explains inhibitory control during childhood: a longitudinal study. Dev Cogn Neurosci. 2014 Jul;9:126-35. doi: 10.1016/j.dcn.2014.02.006. Epub 2014 Feb 27. PMID 24642370